CLINICAL TRIAL: NCT03139175
Title: Association Between Temporomadibular Disorder and Low Back Pain
Brief Title: Association Between TMD and LBP Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Kuei-Chen Lee, Physical therapist, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KLee
Record Dates: First submitted 2017-04-19; First posted 2017-05-03 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Conditions
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- temporomandibular disorder group (Experimental): subjects with TMD and CLBP symptoms undergo balance assessment with Biodex balance system
  Interventions: Device: balance assessment with Biodex balance system
- chronic low back pain group (Active Comparator): subjects only with LBP symptoms undergo balance assessment with Biodex balance system
  Interventions: Device: balance assessment with Biodex balance system
- Normal (Other): subjects without temporomandibular disorder and low back pain symptoms undergo balance assessment with Biodex balance system
  Interventions: Device: balance assessment with Biodex balance system

INTERVENTIONS:
Device: balance assessment with Biodex balance system — All subjects of three groups will be assessed with the evaluation device( balance system).

SUMMARY:
Investigate the relationships between temporomandibular disorder and low back pain

DETAILED DESCRIPTION:
Some patients with chronic low back pain reveal temporomandibular disorder,and others do not. So the aims of my study were to find out the risk factors that contribute to the concurrence of temporomandibular disorder.

ELIGIBILITY:
Inclusion Criteria:

* unilateral LBP for more than 1 year

Exclusion Criteria:

* sensory or neurologic disorders; structural defect of the spine or lower extremities; a history of spine or TMD surgery; recent hip, knee, or ankle pain; any medication that could affect balance; a history of uncorrected visual impairment; and vestibular disorders.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-06 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
balance assesment | only measure the balance performance before the treatment
  The subjects from three groups all receive the balance assessment with the Biodex balance system, and compare the difference.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Chen Lee, MS, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
I can share the conclusions of my research.